CLINICAL TRIAL: NCT06956183
Title: The Effect of Vestibular Exercise Program on Fatigue, Balance and Gait in Patients With Stroke
Brief Title: Effect of Vestibular Exercises on Post-Stroke Fatigue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, ayla fil balkan, associate professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-23056
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Stroke; Vestibular Exercise; Fatigue; Balance; Gait
MeSH Terms: conditions — Stroke; Fatigue

STUDY DESIGN:
Intervention Model Description: Randomized Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Participants in the control group will participate in a one-hour conventional exercise program three times a week for eight weeks.
  Interventions: Other: Control (Standard treatment)
- Vestibular Group (Experimental): In vestibular group (study group) participants in the study group will receive 20 minutes of vestibular training in addition to a 40-minute conventional exercise program, three times a week for eight weeks.
  Interventions: Other: Vestibular exercise

INTERVENTIONS:
Other: Control (Standard treatment) — In control group participants will take one hour conventional physiotherapy including stretching, strengthening, balance and gait exercises in each session.
  Arms: Control group
Other: Vestibular exercise — In vestibular group (study group) participant will take 40 minutes conventional physiotherapy including stretching, strengthening, balance and gait exercises, and 20 minutes vestibular exercises including head and gaze stabilization, occulomotor, head turning and balance exercises in different postures.
  Arms: Vestibular Group

SUMMARY:
The goal of this clinical trial is to search effects of vestibuler exercises on post-stroke fatigue. The main question it aims to answer is:

wer are:

- Do vestibuler excercises decrease post-stroke perceived and physiologic fatigue?

Researchers will compare the effects of vestibuler exercises to conventional rehabilitation to find out the superior one.

Participants will:

* take a one-hour conventional rehabilitation or vestibuler exercise program three times in a week.
* be assessed in terms of fatigue before and after rehabilitation programs.

DETAILED DESCRIPTION:
One of the most common complications after stroke is fatigue. Fatigue prolongs the rehabilitation period and delays recovery. Although medical treatments, exercise programs and activity modifications are recommended to reduce fatigue after stroke, an effective evidence-based treatment method has not yet been developed. Vestibular exercises can improve oculomotor and postural control by trying to provide sensory integration through adaptation and compensatory mechanisms, thus increasing cortical excitability and reducing fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study Being between the ages of 18-65 Having had an anterior circulation stroke at least 6 months ago Being at least stage 3 according to the Functional Ambulation Classification Scoring at least 22 on the Montreal Cognitive Assessment Scale

Exclusion Criteria:

* Having another orthopedic, neurological or other systemic disease that prevents working Having severe aphasia Having a disease other than stroke that causes primary fatigue Using medication that will affect cognitive status Using medication that will affect fatigue

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Fatigue Impact Scale | One week before rehabilitation program and one week after rehabilitation program.
  The Fatigue Impact Scale (FIS) will be used. The FIS, which provides information on the presence and severity of fatigue, asks patients to evaluate 10 physical, 10 cognitive, and 20 psychosocial function-related statements within the scope of their fatigue levels in the last month. Each statement can take a value between 0 and 4. 0 indicates no problem, while 4 indicates the most severe problem. The total scale score varies between 0 and 160. A higher score indicates that the effect of fatigue is greater.
The Fatigue Assessment Scale | One week before rehabilitation program and one week after rehabilitation program.
  The Fatigue Assessment Scale (FAS) consists of 10 items. Responses are given on a five-point Likert scale, with 1 for "never" and 5 for "always". The FAS asks participants to rate how they feel on a daily basis.

SECONDARY OUTCOMES:
Symbol Digit Modalities Test | One week before rehabilitation program and one week after rehabilitation program.
  Physiological mental fatigue will be assessed with the Symbol Digit Modalities Test (SDMT). In the test, 9 numbers are represented by 9 symbols. In the test, participants will be asked to match the symbols given in a mixed manner with the numbers for a period of 180 seconds by looking at the guide. The number of correct answers will be recorded 6 times, every 30 seconds. The difference between the cognitive fatigue value 1. Score and 6. Score will be recorded as the fatigue value.
Six Minutes Walking Test | One week before rehabilitation program and one week after rehabilitation program.
  The assessment of physiological fatigue will be made by calculating the time-dependent change in walking distance with the ambulatory walking index as a result of the 6-minute walking test (6MWT). At the beginning of the test, participants will be instructed to complete "as much distance as possible, aiming to complete at the highest speed". The distances walked per minute and the total distance will be recorded and expressed in meters. In order to measure the decrease in the distance walked from the first minute to all other minutes of the 6-minute walking test, the percentage change in the distance walked will be calculated starting from the second minute. Objective measurement of fatigue will be made by decreasing walking distance between 1 and 6 minutes.

OTHER OUTCOMES:
Fugl Meyer Assessment | One week before rehabilitation program and one week after rehabilitation program.
  Motor functionality will be assessed with the Fugl Meyer Upper Extremity (FMA-UE) and Fugl Meyer Lower Extremity (FMA-LE) scales. FMA-UE is a frequently used assessment tool to assess motor recovery of the upper extremity after stroke. Scoring is as follows; 0= cannot perform, 1= partially perform, 2= fully perform. The total score for upper extremity motor function is 66. FMA-LE is a disease-specific impairment assessment designed to assess motor function, balance, sensory qualities, and joint function in patients after stroke. Scoring is as follows; 0= cannot perform, 1= partially perform, 2= fully perform.
Fullerton Advanced Balance Scale | One week before rehabilitation program and one week after rehabilitation program.
  Fullerton Advanced Balance Scale is a scale developed to evaluate small changes in balance in multiple ways. The highest score that can be obtained from the scale consisting of 10 items scored between 0 and 4 is 40. FAB is a scale that can be applied quickly (∼10-12 min) and does not require space. Its validity and reliability have been shown in stroke patients, and the cut-off score has been determined as 21.5.
Timed Up and Go Test | One week before rehabilitation program and one week after rehabilitation program.
  Timed Up and Go Test; verbal instructions are given to the patient, and the patient is asked to get up from the chair, walk 3 meters as quickly and safely as possible following a line marked on the floor, turn, walk back and sit down. 10 seconds and below; the patient walks independently, the risk of falling is very low. 11-19 seconds; the patient walks independently, the risk of falling is low to moderate. 20-29 seconds; the patient may need help from time to time, the risk of falling is moderate to high. Over 30 seconds, the risk of falling is high and the need for help from time to time
Bertec Force Plate (Balance Check Screener™ BP5050 20x20´´ Bertec Comporation Columbus, OH, USA) | One week before rehabilitation program and one week after rehabilitation program.
  Bertec force plate (Balance Check Screener™ BP5050 20x20´´ Bertec Comporation Columbus, OH, USA) is a three-component balance platform that is based on objectively measuring instantaneous changes in vertical force and pressure center. It consists of a total of 5 tests, including tests for 4 different situations in static stance and a test that includes stability limits. The participant is asked to wait 10 seconds without moving in each situation with eyes open and eyes closed on hard and soft ground. Oscillations are recorded by the device for evaluation during the test.
The GAITRite Gait Analysis System (CIR Systems Inc., Franklin, New Jersey, USA) | One week before rehabilitation program and one week after rehabilitation program.
  The GAITRite Gait Analysis System (CIR Systems Inc., Franklin, New Jersey, USA) will be used to evaluate the participants' gait cycle time, gait speed (cm/s), cadence (step/min), step length (cm), double step length (cm), step width (cm), foot angle (°), support surface (cm), single leg stance time (%GC), and time-distance characteristics of individuals' gait, such as plantar pressure distributions, while they walk at their own pace. The GAITRite system is considered the gold standard in the evaluation of time-distance characteristics of gait (29). The participants' walks will be repeated 3 times and the average of the data related to the gait will be used in the analyses
Functional Gait Assessment | One week before rehabilitation program and one week after rehabilitation program.
  Walking performance and functionality will be assessed with the Functional Gait Assessment (FGA). The FGA is an ambulation-based balance test initially proposed to assess higher-level balance in individuals with vestibular disorders. Although it was developed for use in patients with vestibular pathologies, it has since been used as an outcome measure in a variety of patient populations. The FGA was developed as a modification of the dynamic gait index to increase reliability and reduce the ceiling effect commonly seen with the DGI, with three items added to the 7 items of the dynamic gait index: "walking with narrow-based support," "walking backward," and "walking with eyes closed." Each of the 10 items in the FGA is scored from 0 to 3, with a best score of 30. Validity and reliability have been demonstrated in stroke patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oppenlander K, Utz KS, Reinhart S, Keller I, Kerkhoff G, Schaadt AK. Subliminal galvanic-vestibular stimulation recalibrates the distorted visual and tactile subjective vertical in right-sided stroke. Neuropsychologia. 2015 Jul;74:178-83. doi: 10.1016/j.neuropsychologia.2015.03.004. Epub 2015 Mar 3. PMID 25744870
- [Background] Ghaffari A, Asadi B, Zareian A, Akbarfahimi M, Raissi GR, Fathali Lavasani F. The Effects of Vestibular Rehabilitation on Poststroke Fatigue: A Randomized Controlled Trial Study. Stroke Res Treat. 2022 Aug 31;2022:3155437. doi: 10.1155/2022/3155437. eCollection 2022. PMID 36090743
- [Background] Mitsutake T, Sakamoto M, Ueta K, Oka S, Horikawa E. Effects of vestibular rehabilitation on gait performance in poststroke patients: a pilot randomized controlled trial. Int J Rehabil Res. 2017 Sep;40(3):240-245. doi: 10.1097/MRR.0000000000000234. PMID 28542112
- [Background] Angelaki DE, Klier EM, Snyder LH. A vestibular sensation: probabilistic approaches to spatial perception. Neuron. 2009 Nov 25;64(4):448-61. doi: 10.1016/j.neuron.2009.11.010. PMID 19945388
- [Background] Tramontano M, Bergamini E, Iosa M, Belluscio V, Vannozzi G, Morone G. Vestibular rehabilitation training in patients with subacute stroke: A preliminary randomized controlled trial. NeuroRehabilitation. 2018;43(2):247-254. doi: 10.3233/NRE-182427. PMID 30040765
- [Background] Su Y, Yuki M, Otsuki M. Non-Pharmacological Interventions for Post-Stroke Fatigue: Systematic Review and Network Meta-Analysis. J Clin Med. 2020 Feb 25;9(3):621. doi: 10.3390/jcm9030621. PMID 32106490
- [Background] Paciaroni M, Acciarresi M. Poststroke Fatigue. Stroke. 2019 Jul;50(7):1927-1933. doi: 10.1161/STROKEAHA.119.023552. Epub 2019 Jun 14. No abstract available. PMID 31195940
- [Background] Bernard-Espina J, Beraneck M, Maier MA, Tagliabue M. Multisensory Integration in Stroke Patients: A Theoretical Approach to Reinterpret Upper-Limb Proprioceptive Deficits and Visual Compensation. Front Neurosci. 2021 Apr 7;15:646698. doi: 10.3389/fnins.2021.646698. eCollection 2021. PMID 33897359
- [Background] Oliveira CB, Medeiros IR, Greters MG, Frota NA, Lucato LT, Scaff M, Conforto AB. Abnormal sensory integration affects balance control in hemiparetic patients within the first year after stroke. Clinics (Sao Paulo). 2011;66(12):2043-8. doi: 10.1590/s1807-59322011001200008. PMID 22189728
- [Background] Jang SH, Lee JH. Impact of sensory integration training on balance among stroke patients: sensory integration training on balance among stroke patients. Open Med (Wars). 2016 Aug 13;11(1):330-335. doi: 10.1515/med-2016-0061. eCollection 2016. PMID 28352817
- [Background] Sharony AF, Engel-Yeger B. Sensory Modulation and Participation in Daily Occupations in Stroke Survivors. Can J Occup Ther. 2021 Dec;88(4):375-383. doi: 10.1177/00084174211047372. Epub 2021 Oct 9. PMID 34632801
- [Background] Schambra HM, Sawaki L, Cohen LG. Modulation of excitability of human motor cortex (M1) by 1 Hz transcranial magnetic stimulation of the contralateral M1. Clin Neurophysiol. 2003 Jan;114(1):130-3. doi: 10.1016/s1388-2457(02)00342-5. PMID 12495773
- [Background] Plewnia C, Lotze M, Gerloff C. Disinhibition of the contralateral motor cortex by low-frequency rTMS. Neuroreport. 2003 Mar 24;14(4):609-12. doi: 10.1097/00001756-200303240-00017. PMID 12657896
- [Background] Kluger BM, Krupp LB, Enoka RM. Fatigue and fatigability in neurologic illnesses: proposal for a unified taxonomy. Neurology. 2013 Jan 22;80(4):409-16. doi: 10.1212/WNL.0b013e31827f07be. PMID 23339207
- [Background] Ponchel A, Bombois S, Bordet R, Henon H. Factors Associated with Poststroke Fatigue: A Systematic Review. Stroke Res Treat. 2015;2015:347920. doi: 10.1155/2015/347920. Epub 2015 May 25. PMID 26101691
- [Background] McGeough E, Pollock A, Smith LN, Dennis M, Sharpe M, Lewis S, Mead GE. Interventions for post-stroke fatigue. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD007030. doi: 10.1002/14651858.CD007030.pub2. PMID 19588416
- [Background] Nadarajah M, Goh HT. Post-stroke fatigue: a review on prevalence, correlates, measurement, and management. Top Stroke Rehabil. 2015 Jun;22(3):208-20. doi: 10.1179/1074935714Z.0000000015. Epub 2015 Mar 17. PMID 25779764